CLINICAL TRIAL: NCT07337018
Title: Valutazione Resezioni Oncologiche e Ricostruzione Con Utilizzo di Impianti Protesici in Chirurgia Oncologica Ortopedica (Evaluation of Oncologic Resections and Reconstruction Using Prosthetic Implants in Orthopedic Oncologic Surgery)
Brief Title: Evaluation of Tumor Resection and Reconstruction With Prosthetic Implants
Acronym: RERIO
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 7224
Record Dates: First submitted 2025-12-11; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Bone Tumor
MeSH Terms: conditions — Bone Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No

SUMMARY:
Bone can be the site of primary malignant tumors or, more commonly, secondary lesions. The most frequent primary tumors are osteosarcoma, chondrosarcoma, and Ewing sarcoma, whereas the malignancies that most commonly metastasize to bone include breast, prostate, lung, kidney, and thyroid cancers.

For the treatment of these conditions-and, in some cases, for locally aggressive benign diseases-a surgical approach is often required, which may result in substantial bone loss. Most commercially available prostheses commonly used in orthopedic surgery are not always suitable, either because of the anatomical location of the procedure or the type of resection planned, and thus the extent of the bone defect to be reconstructed. Therefore, specific prosthetic implants designed for oncologic surgery are required.

For this reason, modular prostheses have been developed, allowing reconstruction of bone defects of varying sizes across different anatomical districts. In recent years, the development and use of 3D-printing technology for producing custom-made prostheses has also increased, with the aim of reconstructing bone defects in areas that are difficult to treat and achieving an accurate reproduction of the patient's anatomy. This technology enables reconstruction in a wide range of skeletal sites. Additionally, it allows for preoperative planning on printed anatomical models and opens the possibility of integrating materials with adjuvant-related properties into the prosthetic design, such as photothermal therapy or antimicrobial features.

Although numerous studies on this topic are available in the literature, they frequently involve small patient cohorts. There is therefore a need to expand case series with longer follow-ups to better assess the reliability and effectiveness of these treatment strategies in the development of reconstructive orthopedic oncologic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age between 30 and 70 years;

Diagnosis of primary malignant or locally aggressive benign bone tumors, or secondary bone lesions with a primary diagnosis of breast, lung, prostate, kidney, or thyroid cancer;

Extensive bone loss precluding the use of currently available prostheses or standard surgical techniques;

Use of modular or custom-made prostheses produced with 3D-printing technology; minimum follow-up of 12 months;

(For patients in the retrospective phase) completion of evaluation questionnaires during outpatient follow-ups;

Obtaining Informed Consent, except for deceased patients enrolled in the retrospective phase of the study.

Exclusion Criteria:

Patients with disease spread to other bone segments;

Age <30 years or >70 years;

Patients who have undergone previous surgical procedures on the involved segment;

Follow-up of less than 1 year;

Incomplete clinical or radiological data sets;

Inability to obtain Informed Consent, except for deceased patients enrolled in the retrospective phase of the study

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary or secondary bone tumors treated at the Policlinico A. Gemelli
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Karnofsky Performance Status | From enrollment for at least one year
  Postoperative quality of life and functional status assessed using the Karnofsky Performance Status score.
Musculoskeletal Tumor Society (MSTS) Score | At final follow-up
  Postoperative functional outcome assessed using the Musculoskeletal Tumor Society (MSTS) scoring system.
Quick Disabilities of the Arm, Shoulder and Hand (QuickDASH) Score | From enrollment for at least one year
  Upper-limb functional outcome assessed using the QuickDASH questionnaire in patients with upper extremity involvement
Oxford Knee Score | From enrollment for at least one year
  Knee functional outcome assessed using the Oxford Knee Score in patients with knee involvement
Harris Hip Score | From enrollment for at least one year
  Hip functional outcome assessed using the Harris Hip Score in patients with hip involvement.

SECONDARY OUTCOMES:
Incidence of postoperative complications | From enrollment for at least one year
  Postoperative complications will be assessed through clinical evaluation and review of medical records, supported by imaging and laboratory findings when indicated. Complications include periprosthetic infection, implant loosening, wound dehiscence, dislocation (for implants including an articular component), and periprosthetic fracture. Each complication will be recorded as present or absent according to standard clinical diagnostic criteria

REFERENCES:
- [Background] Sambri A, Zucchini R, Giannini C, Zamparini E, Viale P, Donati DM, De Paolis M. Silver-coated (PorAg(R)) endoprosthesis can be protective against reinfection in the treatment of tumor prostheses infection. Eur J Orthop Surg Traumatol. 2020 Dec;30(8):1345-1353. doi: 10.1007/s00590-020-02705-3. Epub 2020 May 24. PMID 32449080
- [Background] Donati F, Di Giacomo G, D'Adamio S, Ziranu A, Careri S, Rosa M, Maccauro G. Silver-Coated Hip Megaprosthesis in Oncological Limb Savage Surgery. Biomed Res Int. 2016;2016:9079041. doi: 10.1155/2016/9079041. Epub 2016 Aug 23. PMID 27642605
- [Background] Wang X, Liu Y, Zhang M, Zhai D, Wang Y, Zhuang H, Ma B, Qu Y, Yu X, Ma J, Ma H, Yao Q, Wu C. 3D Printing of Black Bioceramic Scaffolds with Micro/Nanostructure for Bone Tumor-Induced Tissue Therapy. Adv Healthc Mater. 2021 Nov;10(21):e2101181. doi: 10.1002/adhm.202101181. Epub 2021 Sep 15. PMID 34523255
- [Background] Zhu C, He M, Sun D, Huang Y, Huang L, Du M, Wang J, Wang J, Li Z, Hu B, Song Y, Li Y, Feng G, Liu L, Zhang L. 3D-Printed Multifunctional Polyetheretherketone Bone Scaffold for Multimodal Treatment of Osteosarcoma and Osteomyelitis. ACS Appl Mater Interfaces. 2021 Oct 13;13(40):47327-47340. doi: 10.1021/acsami.1c10898. Epub 2021 Sep 29. PMID 34587454
- [Background] Girolami M, Boriani S, Bandiera S, Barbanti-Brodano G, Ghermandi R, Terzi S, Tedesco G, Evangelisti G, Pipola V, Gasbarrini A. Biomimetic 3D-printed custom-made prosthesis for anterior column reconstruction in the thoracolumbar spine: a tailored option following en bloc resection for spinal tumors : Preliminary results on a case-series of 13 patients. Eur Spine J. 2018 Dec;27(12):3073-3083. doi: 10.1007/s00586-018-5708-8. Epub 2018 Jul 23. PMID 30039254
- [Background] Liang H, Yang Y, Guo W, Yan L, Tang X, Li D, Qu H, Zang J, Du Z. Elbow hemiarthroplasty with a 3D-printed megaprosthesis for defects of the distal humerus or proximal ulna after tumour resection : a preliminary report. Bone Joint J. 2022 Jun;104-B(6):747-757. doi: 10.1302/0301-620X.104B6.BJJ-2021-1516.R1. PMID 35638204
- [Background] Park JH, Jung HW, Jang WY. The usefulness of a three-dimensional printed segmental scapula prosthesis for recovering shoulder function in a patient with scapula chondrosarcoma: A case report. Medicine (Baltimore). 2021 Feb 26;100(8):e24817. doi: 10.1097/MD.0000000000024817. PMID 33663101
- [Background] Beltrami G, Ristori G, Nucci AM, Galeotti A, Tamburini A, Scoccianti G, Campanacci D, Innocenti M, Capanna R. Custom-Made 3D-Printed Implants as Novel Approach to Reconstructive Surgery after Oncologic Resection in Pediatric Patients. J Clin Med. 2021 Mar 4;10(5):1056. doi: 10.3390/jcm10051056. PMID 33806387
- [Background] Gursan O, Celtik M, Yanik B, Husemoglu RB, Havitcioglu H. Three-Dimensionally-Printed Joint-Preserving Prosthetic Reconstruction of Massive Bone Defects After Malignant Tumor Resection of the Proximal Tibia. Cureus. 2021 Mar 9;13(3):e13784. doi: 10.7759/cureus.13784. PMID 33842159
- [Background] Yang QD, Mu MD, Tao X, Tang KL. Three-dimensional printed talar prosthesis with biological function for giant cell tumor of the talus: A case report and review of the literature. World J Clin Cases. 2021 May 6;9(13):3147-3156. doi: 10.12998/wjcc.v9.i13.3147. PMID 33969102
- [Background] Xu L, Qin H, Cheng Z, Jiang WB, Tan J, Luo X, Huang W. 3D-printed personalised prostheses for bone defect repair and reconstruction following resection of metacarpal giant cell tumours. Ann Transl Med. 2021 Sep;9(18):1421. doi: 10.21037/atm-21-3400. PMID 34733973
- [Background] Chen G, Yin Y, Chen C. Limb-salvage surgery using personalized 3D-printed porous tantalum prosthesis for distal radial osteosarcoma: A case report. Medicine (Baltimore). 2021 Nov 19;100(46):e27899. doi: 10.1097/MD.0000000000027899. PMID 34797342
- [Background] Pu F, Liu J, Shi D, Huang X, Zhang J, Wang B, Wu Q, Zhang Z, Shao Z. Reconstruction With 3D-Printed Prostheses After Sacroiliac Joint Tumor Resection: A Retrospective Case-Control Study. Front Oncol. 2022 Jan 4;11:764938. doi: 10.3389/fonc.2021.764938. eCollection 2021. PMID 35059310
- [Background] Wang S, Luo Y, Zhang Y, Wang Y, Zheng C, Tu C, Zhou Y. Case Report: Reconstruction of Medialis Malleolus (1/4 of the Ankle Joint) After Resection of Distal Tibia Tumor With an Uncemented Three-Dimensional-Printed Prosthesis. Front Surg. 2022 Mar 24;9:844334. doi: 10.3389/fsurg.2022.844334. eCollection 2022. PMID 35402484
- [Background] Park JW, Kang HG. Application of 3-dimensional printing implants for bone tumors. Clin Exp Pediatr. 2022 Oct;65(10):476-482. doi: 10.3345/cep.2021.01326. Epub 2021 Dec 23. PMID 34942688
- [Background] Zhang HR. Application and Development of Megaprostheses in Limb Salvage for Bone Tumors Around the Knee Joint. Cancer Control. 2022 Jan-Dec;29:10732748221099219. doi: 10.1177/10732748221099219. PMID 35499495
- [Background] Thorkildsen J, Strom TA, Strom NJ, Sellevold S, Norum OJ. Megaprosthesis for Metastatic Bone Disease-A Comparative Analysis. Curr Oncol. 2022 May 10;29(5):3460-3471. doi: 10.3390/curroncol29050279. PMID 35621669
- [Background] Denissen JJPM, Koenders N, van Hinte G, Groen F, van der Wees PJ, van der Geest ICM, Dierselhuis EF. Functional outcomes after reverse shoulder megaprosthesis following resection of malignant bone tumor in the proximal humerus: a systematic review and meta-analysis. JSES Int. 2023 Mar 31;7(4):592-600. doi: 10.1016/j.jseint.2023.02.018. eCollection 2023 Jul. PMID 37426912